CLINICAL TRIAL: NCT06503042
Title: A Study to Prospectively Validate Blood Markers Associated With Differences in Efficacy of Neoadjuvant Therapy for Non-small Cell Lung Cancer
Brief Title: A Study to Prospectively Validate Blood Markers Associated With Differences in Efficacy of Neoadjuvant Therapy for NSCLC
Status: Not yet recruiting | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K202407-07
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chemotherapy combined with immunotherapy group: NSCLC patients undergoing neoadjuvant chemotherapy combined with immunotherapy regimens
  Interventions: Drug: Chemotherapy combined with immunotherapy
- Chemotherapy group: NSCLC patients undergoing neoadjuvant chemotherapy regimens
  Interventions: Drug: Chemotherapy only

INTERVENTIONS:
Drug: Chemotherapy combined with immunotherapy — Patients in the chemotherapy combined with immunotherapy group use any chemotherapy drug in combination with any immunotherapy drug. The premise is that the treatment regimen for patients is consistent with the diagnostic and treatment protocols.
  Groups: Chemotherapy combined with immunotherapy group
Drug: Chemotherapy only — Patients in the chemotherapy alone group use any chemotherapy drug. The premise is that the treatment regimen for patients is consistent with the diagnostic and treatment protocols.
  Groups: Chemotherapy group

SUMMARY:
This study utilized a prospective cohort design. It is proposed to analyze the serum of NSCLC patients treated with chemotherapy combined with immunotherapy, and chemotherapy alone, starting from liquid biopsy technique and combining with proteomic methods. By comparing the differences in serum proteins between the two groups of patients before treatment, we will validate the targets related to efficacy and AE events identified in a previous retrospective study, further explore their associations with patients' clinical outcomes and AE events, and establish a clinical prediction model to guide and improve the current treatment of NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must sign the written informed consent form (ICF), and be able to follow the visits and relevant procedures specified in the protocol
2. Cytologically or histologically confirmed primary NSCLC (including adenocarcinoma, squamous cell carcinoma, adenosquamous carcinoma)
3. Have not received any prior systemic anti-tumor therapy or local radiotherapy for NSCLC
4. Have adequate organ and bone marrow function, and the laboratory examination values within 14 days prior to enrollment meet the following requirements (no blood components, cell growth factors, albumin and other intravenous or subcutaneously administered drugs to correct hematological or liver and kidney dysfunction were allowed within the first 14 days of obtaining laboratory tests), as follows:

   ①Hematological function was sufficient, defined as absolute neutrophil count ≥ 1.5 × 109 / L, platelet count ≥ 100 × 109 / L, hemoglobin ≥ 100g / L;

   ②Full liver function, defined as total bilirubin level ≤ 1.5 × ULN, AST and ALT level ≤ 2.5 × ULN, albumin (ALB) ≥ 35g / L;
   * Renal function was sufficient, serum creatinine (Scr) ≤ 1.5 × ULN, creatinine clearance rate (CrCl) ≥ 60mL / min (calculated by Cockcroft / Gault formula) and urine routine test results showed that urinary protein (UPRO) < 2 + or 24-hour urinary protein < 1g;

     * The international normalized ratio (INR) ≤ 1.5 × ULN, and prothrombin time (PT) or activated partial thromboplastin time (APTT) ≤ 1.5 × ULN within 7 days before treatment;
5. For women of childbearing age, urine or serum pregnancy tests were negative for at least seven days prior to the first study drug administration. If the urine pregnancy test is positive, a blood pregnancy test is required;
6. If there is a risk of conception, male and female patients need to use high-efficiency contraception (i.e., the method with an annual failure rate of less than 1 %) and continue until at least 180 days after discontinuation of the trial; Note: If abstinence is the normal lifestyle and preferred contraceptive method of the subjects, abstinence can be accepted as a contraceptive method.

   -

Exclusion Criteria:

1. Pathological examination showed that small cell carcinoma, neuroendocrine carcinoma, sarcoma, lymphoepithelioma-like carcinoma, salivary gland tumor and mesenchymal tumor components
2. Tumor invasion of the diaphragm, mediastinum, heart, pericardium, large blood vessels (such as aorta), esophagus, vertebral body
3. pulmonary sulcus tumor
4. Contralateral lung nodules, it need biopsy if clinically suspected
5. Subjects with confirmed or suspected brain metastases
6. Participation in an interventional clinical study or treatment with another investigational drug or investigational device within 4 weeks prior to enrollment
7. Previous use of anti-PD-1, anti-PD-L1, anti-programmed death receptor ligand 2 (PD-L2) or anti-cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) drugs or any other drugs acting on T cell co-stimulation or immune checkpoint pathways (such as OX40, CD137, etc.) and adoptive cellular immunotherapy
8. Received immunomodulatory drugs (including thymidine, interferon, interleukins, etc.) within the first 4 weeks of enrollment
9. Live attenuated vaccine within the first 4 weeks of enrollment (or plan to receive live attenuated vaccine during the study period). Note: Inactivated seasonal influenza vaccine is permitted, but live attenuated influenza vaccine is not permitted
10. Requires prolonged systemic glucocorticoid use and has received any other form of immunosuppressive therapy within 7 days prior to enrollment Note: Nasal spray, inhalation, or other topical glucocorticoid or physiologic doses of systemic glucocorticoid (≤ 10 mg/day of prednisone or equivalent) are permitted or are used for pretreatment (e.g., for prevention of contrast allergy).
11. History of non-infectious pneumonia requiring glucocorticoid therapy within 1 year prior to enrollment or current interstitial lung disease (≥ grade 2)
12. Active autoimmune disease including, but not limited to, inflammatory bowel disease such as ulcerative colitis or Crohn's disease requiring systemic therapy (e.g., use of disease modifying medications, corticosteroids, or immunosuppressive drugs) within the 2 years prior to enrollment Diverticulitis, celiac disease, systemic lupus erythematosus, sarcoidosis-like or Wegener's syndrome (granulomatous polyangiitis), Graves' disease, rheumatoid arthritis, multiple sclerosis, vasculitis, glomerulonephritis rheumatoid arthritis, multiple sclerosis, vasculitis, glomerulonephritis, antiphospholipid syndrome, pituitary gland inflammation, and uveitis. Replacement therapies (e.g., thyroxine, insulin, or physiologic doses of corticosteroids for adrenal or pituitary dysfunction) are not considered systemic therapy. Patients with positive autoimmune antibodies will be enrolled only after evaluation by the investigator to confirm that there are no autoimmune diseases requiring systemic therapy.
13. Primary immunodeficiency diseases
14. Pre-existing or current myocarditis
15. incomplete recovery from toxicity and/or complications resulting from any intervention prior to enrollment (> grade 1 or not recovered to baseline levels)
16. Peripheral neuropathy ≥ grade 2
17. Hereditary predisposition to bleeding or coagulation disorders, or history of thrombosis: Any arterial thrombosis, embolism, or ischemia such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, or pulmonary embolism within 6 months prior to enrollment. History of deep vein thrombosis or any other serious thromboembolism within 3 months prior to enrollment (implantable venous access ports or catheter-derived thrombosis or superficial vein thrombosis are not considered thromboembolism).
18. Subjects with non-squamous NSCLC who are unable or unwilling to supplement with folic acid or vitamin B12
19. Any unstable systemic disease or complication, including but not limited to 1) active infection (requiring anti-infective medications or systemic anti-infective medications within one week prior to randomization); 2) congestive heart failure [New York Heart Association, NYHA ≥ Class II]; 3) severe cardiac arrhythmia, hepatic, renal, or metabolic disorders requiring medication; 4) untreated atherosclerotic heart disease of the coronary arteries; 5) history of gastrointestinal perforation and/or fistulae (5) History of gastrointestinal perforation and/or fistula; (6) History of intestinal obstruction, extensive bowel resection or chronic diarrhea within the past 6 months.
20. Solid organ or blood system transplantation.
21. Have a history of HIV infection (HIV1/2 antibody positive), active syphilis
22. Tuberculosis, which is active or requires medical intervention at this stage, including but not limited to pulmonary tuberculosis
23. Active Hepatitis B Subjects with hepatitis B who met the following criteria met the inclusion criteria: HBsAg (+) or HBcAb (+), HBV viral load < 2000 copies/ml or < 200 IU/ml or lower than the detection limit HBsAg Subjects with anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load (-) do not need to receive prophylactic anti-HBV treatment, but need to closely monitor whether the virus is reactivated
24. Active hepatitis C (HCV antibody positive and HCV-RNA level above the detection limit)
25. patients with malignancies other than diagnosed NSCLC within the first 5 years of enrollment, with the exception of fully treated carcinoma in situ of the cervix, basal cell or squamous cell skin cancer, localized prostate cancer after radical surgery, ductal carcinoma in situ after radical surgery, and papillary thyroid cancer after radical therapy
26. Hypersensitivity to the active ingredient(s) and/or any excipient(s) of the chemotherapeutic or immunotherapeutic regimen.
27. Pregnant or lactating women or women who intend to become pregnant or breastfeed during the study period
28. Subjects with mental illness or substance abuse that may interfere with compliance with trial requirements and a history of alcohol abuse
29. non-malignant tumors due to localized or systemic disease, or secondary reactions to cancer, that can lead to higher medical risk and/or uncertainty in survival assessment, in the opinion of the investigator, caused by the subject having a medical history, disease, treatment, or laboratory abnormality that may interfere with the results of the trial, that prevents the subject from participating in the study in its entirety, or in the opinion of the investigator, that the subject will not receive optimal benefit from the study.

    -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with non-small cell lung cancer undergoing neoadjuvant chemotherapy combined with immunotherapy or neoadjuvant chemotherapy at the Thoracic Surgery Department of Tang Du Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 4 months
  rate of pathological complete response
MPR rate | 4 months
  rate of major pathologic response

SECONDARY OUTCOMES:
AE | 4 months
  Adverse Event

IPD SHARING:
Plan to Share IPD: No